CLINICAL TRIAL: NCT04763538
Title: Quality and Outcome Measurements of Urological Patients
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Hospital Centre Biel/Bienne (Other)
Responsible Party: Sponsor
Other Study IDs: ID 2020-02852
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Urologic Diseases
MeSH Terms: conditions — Urologic Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of care — Patients are treated according to the standard of care for each individual disease.

SUMMARY:
Prospectively, all available parameters of urologic patients treated at the study sites will be acquired and stored in multilayered databases. Upon a given samples size, neuronal networks will be trained to define clinical endpoints. Beside uro-oncological patients also patients with other urological diseases will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at the study sites, signed informed consent

Exclusion Criteria:

* No consent to record medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Entire patient population that is treated at the study sites
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease specific primary endpoint | 4-5 years
  Neuronal networks will be trained to define the respective endpoints for the diseases

CONTACTS AND LOCATIONS:
Overall Officials: Roland Seiler, Prof., Study Chair — Department of Urology, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Roland Seiler, Biel
  - Department of Urology, Hospital Center Biel, Biel

IPD SHARING:
Plan to Share IPD: No
In this trial, the investigators will record complete patient data in our multilayered databases. They will be used to train neuronal networks. Latter can be shared with researchers, the multilayered databases will not be shared.